CLINICAL TRIAL: NCT06520358
Title: Acute Intermittent Hypoxia to Improve Airway Protection in Chronic Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB202301156
Record Dates: First submitted 2024-07-19; First posted 2024-07-25 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2024-11

CONDITIONS: Traumatic Brain Injury
Keywords: acute intermittent hypoxia; rehabilitation; airway protection; dysphagia
MeSH Terms: conditions — Brain Injuries, Traumatic; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: The pilot study will utilize a double-blind, placebo-controlled, randomized-order, repeated-measures, cross-over experimental design
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and assessors will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AIH + TST (Active Comparator): Participants will complete a 5-day intervention blocks where they receive daily AIH followed by task specific airway protection training 60 minutes after the AIH exposure. Each exposure involves a 1-minute delivery of low oxygen (9-11% inspired O2), followed by a 1.5-min interval of room air breathing (21% O2). This method of waiting 45-60 minutes after the delivery of AIH and prior to engaging in task-specific training/rehabilitation enables sufficient time to increase brain derived neurotrophic factor (BDNF) following AIH, thereby augmenting the impact of task-specific training.
  Interventions: Other: Acute Intermittent Hypoxia (AIH); Behavioral: Task specific Airway Protection Training
- Sham AIH + TST (Sham Comparator): Participants will complete a 5-day intervention blocks where they receive sham AIH followed by task specific airway protection training 60 minutes after the AIH sham exposure. Sham AIH will be delivered using methods identical to AIH, except a normoxic gas mixture (~21% O2) will be delivered. The gas mixture with normoxic air will effectively serve as a sham.
  Interventions: Behavioral: Task specific Airway Protection Training; Other: Sham AIH

INTERVENTIONS:
Other: Acute Intermittent Hypoxia (AIH) — Acute intermittent hypoxia refers to brief (acute), repetitive (intermittent) episodes of breathing oxygen-deprived air (hypoxia) alternating with breathing ambient room air.
  Arms: AIH + TST
Behavioral: Task specific Airway Protection Training — The vLVC maneuver involves training participants to volitionally prolong closure of the laryngeal vestibule during swallowing, beginning with swallow onset and sustaining closure for at least 2 seconds.
  Other Names: volitional laryngeal vestibule closure (vLVC) training
Other: Sham AIH — Sham AIH will be delivered using methods identical to AIH, except a normoxic gas mixture (~21% O2) will be delivered. The gas mixture with normoxic air will effectively serve as a sham.
  Arms: Sham AIH + TST

SUMMARY:
Acute intermittent hypoxia (AIH) involves 1-2min of breathing low oxygen air to stimulate neuroplasticity. Animal and human studies show that AIH improves motor function after neural injury, particularly when paired with task-specific training. Using a double blind cross-over study we will test whether AIH and task-specific airway protection training improves airway protection more than training alone in individuals with chronic mild-moderate traumatic brain injury (TBI).

DETAILED DESCRIPTION:
Recent studies have found that acute intermittent hypoxia (AIH)-or repetitive exposure to brief episodes of low inspired oxygen--is a promising new strategy that can help restore motor function by promoting neuroplasticity throughout the central nervous system (CNS). Both rodent and human studies show that motor function is further enhanced when AIH is paired with task-specific training/rehabilitation (TST). Therefore, this study will investigate the therapeutic potential of combining AIH with a task-specific airway protection training. We propose that the combined use of AIH + TST will enhance the magnitude and duration of TST training alone in individuals with chronic traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 21-80 years
* A mild to moderate traumatic brain injury (TBI) confirmed by medical records
* A Glasgow Coma Scale score between 9-15
* Able to consent independently
* Women of child-bearing age must be comfortable confirming a negative pregnancy prior to participating in the study

Exclusion Criteria:

* Other neurological diagnoses or a diagnosis of a severe psychiatric disorder
* Severe aphasia preventing a participant from understanding the protocol and consent form
* Pre-existing hypoxic pulmonary disease
* History of obstructive lung diseases such as chronic obstructive pulmonary disease (COPD) or significant asthma)
* Severe hypertension (>160/100)
* History of head and neck cancer
* Allergy to barium sulfate
* Ischemic cardiac disease

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Duration of laryngeal vestibule closure (dLVC) | Pre-intervention, 1 day after intervention block and 1-week post intervention
  Time in (msec) the laryngeal vestibule stays closed during a swallow
Time to laryngeal vestibule closure (Time-to-LVC) | Pre-intervention, 1 day after intervention block and 1-week post intervention
  Time in (msec) it takes to close the laryngeal vestibule after swallow initiation

SECONDARY OUTCOMES:
Penetration-Aspiration Scale Scores | Pre-intervention, 1 day after intervention block and 1-week post intervention
  The penetration-aspiration scale (PAS) will be used to assess penetration or aspiration; the PAS is an 8-point scale that ranges from 1 (no penetration/aspiration) to 8 (aspiration with no cough response).

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Z Vose, Ph.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vose AK, Welch JF, Nair J, Dale EA, Fox EJ, Muir GD, Trumbower RD, Mitchell GS. Therapeutic acute intermittent hypoxia: A translational roadmap for spinal cord injury and neuromuscular disease. Exp Neurol. 2022 Jan;347:113891. doi: 10.1016/j.expneurol.2021.113891. Epub 2021 Oct 9. PMID 34637802
- [Background] Welch JF, Sutor TW, Vose AK, Perim RR, Fox EJ, Mitchell GS. Synergy between Acute Intermittent Hypoxia and Task-Specific Training. Exerc Sport Sci Rev. 2020 Jul;48(3):125-132. doi: 10.1249/JES.0000000000000222. PMID 32412926
- [Background] Vose A, Humbert I. "Hidden in Plain Sight": A Descriptive Review of Laryngeal Vestibule Closure. Dysphagia. 2019 Jun;34(3):281-289. doi: 10.1007/s00455-018-9928-1. Epub 2018 Jul 30. PMID 30062547